CLINICAL TRIAL: NCT04099368
Title: Music Appreciation After Cochlear Implantation
Acronym: MACI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Ohio State University (Other); University of California, Merced (Other)
Responsible Party: Principal Investigator, Raymond Goldsworthy, Associate Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01DC018701-01 (NIH)
Record Dates: First submitted 2019-09-17; First posted 2019-09-23 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-06

CONDITIONS: Hearing Loss; Cochlear Implants
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Auditory (Experimental): Group receives training on listening to musical pitch differences between sounds as the first component of a crossover trial. The intervention is the listening exercises. Exercises are completed daily as 30-minute sessions for 4 weeks. Hearing assessment outcomes of speech comprehension in background noise and of musical pitch sensitivity are conducted at baseline and at midpoint and endpoint.
  Interventions: Behavioral: Musical pitch training
- Visual (Active Comparator): Group receives training on visual differences between objects on a computer screen as the first component of a crossover trial. This is a control measure for the auditory training exercises. Exercises are completed daily as 30-minute sessions for 4 weeks. Hearing assessment outcomes of speech comprehension in background noise and of musical pitch sensitivity are conducted at baseline and at midpoint and endpoint.
  Interventions: Behavioral: Musical pitch training

INTERVENTIONS:
Behavioral: Musical pitch training — Crossover design with one group receiving musical training as rehabilitation, second group receiving visual training first as a control rehabilitation.
  Other Names: Auditory rehabilitation

SUMMARY:
This project aims to characterize the emergence of music appreciation in people who have suffered hearing loss and have been provided with partial restoration of hearing through cochlear implantation. Music appreciation is complex and transverses multiple domains including hearing acuity, speech and language acquisition, and quality of life. By studying these relationships in people who have been given partial hearing restoration, the investigators will clarify the role of music for promoting recovery from debilitating loss.

DETAILED DESCRIPTION:
Cochlear implants are medical devices that restore a remarkable degree of hearing to people who would otherwise be profoundly deaf. These devices generally restore enough hearing that recipients can understand spoken speech even in noisy environments. However, most recipients express dissatisfaction with music. This proposal centers on understanding the challenges that implant users face and the strategies that they adopt as they learn to appreciate music with this new way of hearing.

The proposed research is organized into three aims:

Aim 1: Characterize music appreciation after cochlear implantation. The proposed research balances qualitative and quantitative methods to examine the emergence of music appreciation after cochlear implantation. Qualitative methods will include semi-structured interviews and focus groups designed to clarify the obstacles that implant users face as they learn to appreciate music with their new sense of hearing. Quantitative methods include surveys of music appreciation and quality of life, and auditory assessments of music and speech perception. The primary hypothesis is that music appreciation is predictive of key domains of quality of life including positive affect and well-being, and satisfaction with social roles and activities.

Aim 2: Determine if pitch training improves cochlear implant speech comprehension. The proposed research tests for a causal relationship between pitch salience and key features of speech perception including talker discrimination, prosody detection, and speech recognition in competing speech. Cochlear implant users and their normal-hearing peers will take part in a crossover study to determine if pitch training improves aspects of music and speech perception compared to a visual task used as a control. The primary hypothesis is that pitch training will improve speech comprehension for cochlear implant users, but not for their normal-hearing peers.

Aim 3: Test the limits of pitch coding in cochlear implants. The proposed research bypasses conventional sound processing to study the salience of pitch provided by electrode location and stimulation rate. These two stimulation cues are the primary cues for providing a sense of pitch to cochlear implant users. New research has shown that implant users are able to learn to use this information to hear pitch with better resolution far better than previously thought. The primary hypothesis is that cochlear implant users have a latent ability to hear pitch associated with stimulation rate, but that they require experience to learn how to hear this new information.

In each aim, psychophysical methods are combined with measures of EEG and near-infrared spectroscopy. The results will establish the importance of music training for improving cochlear implant outcomes, both in terms of hearing abilities and quality of life. The results will lead to changes in how music is encoded into implant stimulation, providing better outcomes for recipients. More generally, this project will shape understanding of neural coding of music and its role in social adjustment following traumatic experiences.

ELIGIBILITY:
Inclusion Criteria:

* Teenage and adult cochlear implant users

Exclusion Criteria:

* Children younger than 13

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Pitch Discrimination measured using Psychophysical Procedures | Measure collected at 0, 4, and 8 week mark to examine change in discrimination thresholds.
  Change in auditory resolution of fundamental frequency is measured using psychophysical procedures.

SECONDARY OUTCOMES:
Change in Speech Recognition Thresholds measured using Psychophysical Procedures | Measure collected at 0, 4, and 8 week mark to examine change in speech recognition thresholds.
  Speech recognition thresholds measured using adaptive procedures for speech recognition in different types of background noise.

CONTACTS AND LOCATIONS:
Locations (1):
- Keck School of Medicine of USC, Los Angeles, California, United States